CLINICAL TRIAL: NCT01507584
Title: The Effects of the Water Drinking Test on Intraocular Pressure of Glaucoma Patients Undergoing 24 Hour Continuous Monitoring With the SENSIMED Triggerfish
Brief Title: The Effects of the Water Drinking Test on Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 110903
Record Dates: First submitted 2011-09-01; First posted 2012-01-11 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prostaglandin Analogue (Active Comparator): WDT protocol Visit 1 - (WDT after washout) 20 Visit 2 - (WDT with treatment) 20 Visit 3 - (WDT with PGA or BB add-on) 20 (PGA + BB)
  Interventions: Device: SENSIMED Triggerfish
- Carbonic Anhydrase Inhibitor (Active Comparator): WDT protocol Visit 1 - (WDT after washout) 20 Visit 2 - (WDT with treatment) 20 Visit 3 - (WDT with PGA or BB add-on) 20 (CAI+ BB)
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Comparison of fluctuation of Intraocular pressures with different class of drugs
  Other Names: bimatoprost (Lumigan); brinzolamide (azopt)

SUMMARY:
This clinical trial is designed to investigate the efficacy profile of the SENSIMED Triggerfish® during 24-hour IOP monitoring in patients with glaucoma or ocular hypertension, done three times at monthly intervals under different therapeutic regimen. This trial will also evaluate the efficacy of SENSIMED Triggerfish® to detect changes in intraocular pressure (IOP) after the water drinking test (WDT) will be investigated.

DETAILED DESCRIPTION:
The investigation will recruit male and female patients 18-80 years old and diagnosed with glaucoma or ocular hypertension requiring hypotensive ocular treatment. Up to 100 subjects will be enrolled in the study to ensure a minimum of 80 completing three IOP fluctuation monitoring sessions. Patients will be considered enrolled in the study upon signature of informed consent. A screening visit and three 26-hour IOP fluctuation monitoring sessions are planned for each patient. IOP monitoring sessions will be carried out in ambulatory mode at 4 week intervals (plus/minus 7 days). All subjects will be monitored during the same period of the day (± 1hr). The expected duration of participation for each patient is of 3.5 days over three to four months. Patients will be recruited over a 16-month period. The total expected study duration is 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to comply with the study procedures
* 18-80 years old
* Subjects diagnosed with glaucoma, based on presence of repeatable visual field loss and/or glaucomatous optic neuropathy based on masked review of optic disc stereophotographs and under ocular hypotensive treatment, or diagnosed with ocular hypertension, with an IOP of > 22 mmHg at the screening visit and under ocular hypotensive treatment.
* Subject has consented to be in the trial
* Visual acuity of 20/80 or better
* Ability to understand the character and individual consequences of the study
* For women of childbearing potential, adequate contraception
* Stable anti-hypertensive treatment regimen 4 weeks prior to the screening visit and throughout the study.

Exclusion criteria

* Subjects with chronic kidney failure and chronic hear disease
* Subjects with contraindications for wearing contact lenses
* Severe dry eye syndrome
* Keratoconus or other corneal abnormality
* Conjunctival or intraocular inflammation
* Eye surgery prior to and throughout the study, except prior uncomplicated cataract surgery and laser a minimum of 3 months prior to the screening visit.
* Full frame metal glasses during SENSIMED Triggerfish® monitoring
* Known hypersensitivity to silicone, plaster or ocular anesthesia (proparacaine)
* Pregnancy and lactation
* Simultaneous participation in other clinical studies
* No patient will be allowed to participate in this trial more than once

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-08; Primary Completion 2013-04-30 (Actual); Study Completion 2013-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaweh Mansouri, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Hamilton Glaucoma Center, UCSD, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has left the institution and the study data can not be located. Multiple attempts where made to reach the study team, so there are no results to report.
Period: Overall Study
Arm/Group | ALL PARTICIPANTS
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and the study data can not be located. Multiple attempts where made to reach the study team, so there are no results to report.
Arm/Group | ALL PARTICIPANTS
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: 24-hour IOP Patterns
Description: Assess IOP patterns between day and night time and changes after the WDT.
Time Frame: 24-hour
Population: as for baseline characteristics
Arm/Group | ALL PARTICIPANTS
Number analyzed (Participants) | 0

2. Primary Outcome: Intraocular Pressure
Description: IOP monitoring sessions will be carried out in ambulatory mode at 4 week intervals (plus/minus 7 days)
Time Frame: 24-hours
Population: as for baseline characteristics
Arm/Group | ALL PARTICIPANTS
Number analyzed (Participants) | 0

3. Secondary Outcome: Ocular Adverse Events
Description: appearance of any device- or non-device-related ocular adverse events
Time Frame: 24-hours
Population: as for baseline characteristics
Arm/Group | ALL PARTICIPANTS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI has left the institution and the study data can not be located. Multiple attempts where made to reach the study team, so there are no results to report.
Arm/Group | ALL PARTICIPANTS
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The PI has left the institution and the study data can not be located. Multiple attempts where made to reach the study team, so there are no results to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes